CLINICAL TRIAL: NCT04474951
Title: Food Supplements to Control Signs and Symptoms Induced by Cancer Therapies
Brief Title: Food Supplements Based on Nettle and Peppermint to Control Signs and Symptoms Induced by Cancer Therapies
Acronym: GALENO 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Claudio Zamagni MD, MD Medical Oncologist, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GALENO 1
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: breast cancer; ovarian cancer; stinging nettle; peppermint; anemia; fatigue; nausea
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Anemia; Fatigue; Nausea | interventions — stinging nettle lectin; peppermint oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anemia (Experimental): Metastatic patients with grade 1 anemia and on treatment with anti-CDK 4/6 or PARP Inhibitors (10 patients) or on adjuvant therapy with hormonal therapy (10 patients) will be enrolled. The control of the event will be evaluated during treatment with 40 drops TID of Stinging Nettle Fluid Extract; hemoglobin levels will be assessed every 4 weeks for a maximum period of 6 months.
  Interventions: Dietary Supplement: Stinging Nettle
- Fatigue (Experimental): Patients on treatment with Epirubicin and Cyclophosphamide or Carboplatin and Taxane and showing fatigue not associated to anemia or with anemia grade 1 (10 patients) or associated to anemia grade 2 (10 patients) will be enrolled. The control of the event will be evaluated during treatment with 40 drops TID of Stinging Nettle Fluid Extract; the assessment of fatigue will be performed at every chemotherapy cycle, for a maximum period of 6 months.
  Interventions: Dietary Supplement: Stinging Nettle
- Nausea (Experimental): 20 patients on treatment with Epirubicin and Cyclophosphamide or Carboplatin and Taxane and showing nausea of any grade (without vomiting) will be enrolled. The control of the event will be evaluated during treatment with 40 drops TID of Peppermint Fluid Extract, associated to antiemetic therapy prescribed as per clinical practice; the assessment of nausea will be performed at every chemotherapy cycle, for a maximum period of 6 months.
  Interventions: Dietary Supplement: Peppermint

INTERVENTIONS:
Dietary Supplement: Stinging Nettle — Eligible patients will take 40 drops TID of Fluid Extract of Stinging Nettle for control of anemia.
  Arms: Anemia
Dietary Supplement: Stinging Nettle — Eligible patients will take 40 drops TID of Fluid Extract of Stinging Nettle for control of fatigue.
  Arms: Fatigue
Dietary Supplement: Peppermint — Eligible patients will take 40 drops TID of Fluid Extract of Peppermint for control of nausea.
  Arms: Nausea

SUMMARY:
The main purpose of this study is to evaluate the impact of food supplements (herbal remedies) on sign and symptoms induced by cancer therapies: Nettle will be administered for improvement of anemia and fatigue; Peppermint will be administered for improvement of nausea. Secondary aims of the trial are to evaluate the impact of these supplements on the quality of life and to evaluate their tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years
* Karnofsky Performance Scale (KPS) ≥ 90%
* Breast or Gynecological cancer
* Informed consent signed before every procedure study specific, on day 1 of therapy cycle
* Inclusion Criteria Arm 1: presence of grade 1 anemia as per CTCAE 4.0 criteria; patients on treatment with anti-CDK 4/6 or PARP Inhibitors or in adjuvant therapy with hormone therapy
* Inclusion Criteria Arm 2: presence of fatigue of any grade; patients on treatment with Epirubicin and Cyclophosphamide or Carboplatin and Taxane
* Inclusion Criteria Arm 3: presence of nausea of any grade, without vomiting; patients on treatment with Epirubicin and Cyclophosphamide or Carboplatin and Taxane

Exclusion Criteria:

* Arm 1, 2 and 3: Previous intake of food supplements within 4 weeks from the enrollment
* Arm 2: patients with evidence of anxiety or anxious-depressive syndrome; Clinical hypothyroidism not compensated by replacement therapy; Persistent insomnia
* Arm 3: patients with evidence of anxiety or anxious-depressive syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Anemia | Patients will be followed from date of enrollment for a maximum period of 6 months. Hemoglobin levels monitoring performed for a maximum period of 6 months or until the worsening of anemia (Hb<10 g/dL).
  Assessment of hemoglobin levels every 4 weeks.
Fatigue | Patients will be followed from date of enrollment for a maximum period of 6 months.
  Evaluation of fatigue with questionnaire "Brief Fatigue Inventory" - BFI, completed by the patients at day 1 of every cycle of chemotherapy.
Nausea | Patients will be followed from date of enrollment for a maximum period of 6 months.
  Evaluation of nausea with questionnaire "Multinational Association of Supportive Care in Cancer" - MAT, completed by the patients at day 2 and day 5 of every cycle of chemotherapy.

SECONDARY OUTCOMES:
Quality of life level: questionnaire | Patients will be followed from date of enrollment for a maximum period of 6 months.
  Evaluation of quality of life with questionnaire EQ-5D, completed at day 1 of every cycle of chemotherapy by patients enrolled in the three arms.
Tolerability of food supplements | Patients will be followed from date of enrollment for a maximum period of 6 months.
  Evaluation of tolerability of food supplements through registration of adverse events at each patient visit.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zamagni, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi SSD Oncologia Medica Addarii
Locations (1):
- Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tayarani-Najaran Z, Talasaz-Firoozi E, Nasiri R, Jalali N, Hassanzadeh M. Antiemetic activity of volatile oil from Mentha spicata and Mentha x piperita in chemotherapy-induced nausea and vomiting. Ecancermedicalscience. 2013;7:290. doi: 10.3332/ecancer.2013.290. Epub 2013 Jan 31. PMID 23390455
- [Background] Rutto LK, Xu Y, Ramirez E, Brandt M. Mineral Properties and Dietary Value of Raw and Processed Stinging Nettle (Urtica dioica L.). Int J Food Sci. 2013;2013:857120. doi: 10.1155/2013/857120. Epub 2013 May 16. PMID 26904610
- [Background] Meral I, Kanter M. Effects of Nigella sativa L. and Urtica dioica L. on selected mineral status and hematological values in CCl4-treated rats. Biol Trace Elem Res. 2003 Winter;96(1-3):263-70. doi: 10.1385/BTER:96:1-3:263. PMID 14716106